CLINICAL TRIAL: NCT05513495
Title: The Effect of Drip Versus Intermittent Feeding on Splanchnic Oxygenation in Preterm Infants With Intrauterine Growth Retardation: A Prospective Randomized Trial
Brief Title: The Effect of Neonatal Feeding Modalities on Splanchnic Oxygenation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ozge Surmeli Onay (Other)
Collaborators: Eskisehir Osmangazi University (Other)
Responsible Party: Sponsor-Investigator, Ozge Surmeli Onay, MD, Associate Professor, Section of Neonatology, Department of Pediatrics Faculty of Medicine, Eskisehir Osmangazi University
Organization: Eskisehir Osmangazi University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: EskisehirOU-OSOnay-1
Record Dates: First submitted 2022-08-22; First posted 2022-08-24 (Actual); Last update posted 2022-08-24 (Actual); Status verified 2022-08

CONDITIONS: Intrauterine Growth Retardation; Feeding Patterns; Splanchnic Hypoperfusion
Keywords: fetal superior mesenteric artery; Intrauterine Growth Retardation; drip feeding; intermittent feeding; regional splanchnic saturation; umbilical catheter
MeSH Terms: conditions — Fetal Growth Retardation; Feeding Behavior

STUDY DESIGN:
Intervention Model Description: A single-center, prospective, randomized trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Drip Group (Active Comparator): Each infant received the same amount of feed via continuous administration for 3 hours, and subsequent feeding resumed 1 hour after the end of continuous feeding. All of the infants were fed through an orogastric tube that was attached to a syringe infusion pump for continuous feeding. Once a full enteral feed of 120 mL/kg/day was achieved, the drip feeding was stopped.
  Interventions: Other: The effect of drip versus intermittent feeding on splanchnic oxygenation
- Intermittent Group (Active Comparator): Every 3 hours (×8/day), each infant received a 10-minute gravity bolus of milk/preterm formula via orogastric tube.
  Interventions: Other: The effect of drip versus intermittent feeding on splanchnic oxygenation

INTERVENTIONS:
Other: The effect of drip versus intermittent feeding on splanchnic oxygenation — After preterm delivery the infants were randomly assigned to one of two feeding modalities: drip (3-hour continuous) or intermittent (bolus in 10 minutes).

SUMMARY:
OBJECTIVES: The main purpose of this study was to evaluate the impact of drip versus intermittent feeding on splanchnic oxygenation in preterm infants with intrauterine growth restriction (IUGR). The second objective was to assess the relationship between fetal splanchnic circulation parameters and splanchnic oxygenation during the first week of life.

METHODS: A single-center, prospective, randomized study with 51 fetuses/infants was conducted. Fetal Doppler measurements including umbilical artery, middle cerebral artery, and superior mesenteric artery (SMA) were recorded in IUGR fetuses. After preterm delivery the infants were randomly assigned to one of two feeding modalities: drip (3-hour continuous) or intermittent (bolus in 10 minutes). Continuous regional splanchnic saturation (rSO2S) monitoring was carried out during first week of life, simultaneously with continuous oxygen arterial saturation (SaO2) monitoring and the infants' fractional oxygen extractions (FOE) were calculated. These parameters were evaluated as means on a daily basis for the first week of life, as well as pre-prandial and post-prandial measurements on the seventh day.

RESULTS: Fetal Doppler flow velocimetry disturbances were present in 72.5% of the study cohort. The Drip (26 infants) and Intermittent (25 infants) groups were similar in demographic and clinical characteristics, as well as the prevalence of feeding intolerance and necrotizing enterocolitis. During the first week of life, there was no difference in daily mean rSO2S and FOE values between the Drip and Intermittent groups, whereas unfed infants had mostly lower rSO2S values. Pre-prandial and post-prandial rSO2S values remained stable in both groups. Also, no association was detected between fetal splanchnic circulation parameters and neonatal splanchnic oxygenation. RSO2S values were strongly correlated to gestational age and birth weight. During the whole week, except for the first two days, infants with umbilical catheters had significantly lower rSO2S values than infants without.

CONCLUSIONS: Our data suggests that the key factor in splanchnic oxygenation is feeding, not the feeding modality. In addition, the umbilical vein catheter had a negative impact on splanchnic oxygenation.

DETAILED DESCRIPTION:
Study design This single-center prospective randomized study was conducted in a university hospital between 1 January 2019-1 October 2021. This work has been supported by Eskisehir Osmangazi University Scientific Research Projects Coordination Unit under grant number 61690618-604.99-E.61140. This study was conducted in conformity with the principles and regulations of the Helsinki Declaration. The Institutional Ethics Committee approved the study (No: 80558721-050.99-E.105607) and informed consent forms were received from all parents/legal guardians of each fetus/infant before inclusion in the study.

Study Cohort The inclusion criteria were that the parents agreed to participate in the study and that Doppler measurements could be performed in fetuses with IUGR and following preterm birth (GA<37 weeks) with no enteral nutrition prior to enrolment. The infants with chromosomal or major congenital abnormalities that may influence the ability to monitor the splanchnic bed (congenital heart defects, abdominal wall defects, or congenital diaphragmatic hernia), inherited metabolic diseases, hydrops fetalis, TORCH infection, multiorgan failure, infants with spontaneous intestinal perforation, infants with skin lesions at the site of sensor placement and infants who were hospitalized shorter than 7 days because of discharge or death were excluded from the study.

ELIGIBILITY:
Inclusion Criteria:

* Doppler measurements must be performed in fetuses with IUGR
* Preterm infants (GA<37 weeks) with IUGR who were evaluated by Doppler ultrasound were eligible for the study
* These preterm infants must have no enteral nutrition prior to enrolment.

Exclusion Criteria:

* Chromosomal or major congenital abnormalities that may influence the ability to monitor the splanchnic bed (congenital heart defects, abdominal wall defects, or congenital diaphragmatic hernia)
* Inherited metabolic diseases
* Hydrops fetalis
* TORCH infection
* Multiorgan failure
* Infants with spontaneous intestinal perforation
* Infants with skin lesions at the site of sensor placement
* Infants who were hospitalized for shorter than 7 days because of discharge or death

Ages: 1 Minute to 3 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 51 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2021-12-01 (Actual); Study Completion 2021-12-01 (Actual)

PRIMARY OUTCOMES:
Fetal SMA Doppler measurements | The last ultrasound study within 48 hours prior delivery was used for analysis.
  Antenatal SMA doppler measurements such as pulsatility index
Daily mean rSO2S&FOE during the first week of life | Continuous rSO2S monitoring was carried out during first week of life.
  Splanchnic saturation and fractional tissue oxygen extractions during the first week of life
Pre-prandial and post-prandial rSO2S&FOE | During seventh day of life, the machine's marking button was pressed when the feeding began (09:00 am and 21:00 pm feeding practices were evaluated for each infant).
  Splanchnic saturation and fractional tissue oxygen extractions at the 7th day of life related to feeding modalities (drip vs intermittent feeding).
The incidence of feeding intolerance, necrotising enterocolitis and time to full enteral feeding | From admission to discharge
  These outcome parameters were evaluated during neonatal intensive care stay

SECONDARY OUTCOMES:
The relationship between fetal splanchnic circulation parameters and neonatal splanchnic oxygenation. | Perinatal period (from 48 hours before delivery to first week of life)
  The relation between fetal SMA doppler parameters and regional splanchnic saturation measurements

CONTACTS AND LOCATIONS:
Overall Officials: Ozge Surmeli Onay, Principal Investigator — Eskisehir Osmangazi University
Locations (1):
- Ozge Surmeli Onay, Eskişehir, Turkey (Türkiye)

REFERENCES:
- [Derived] Surmeli Onay O, Velipasaoglu M, Tutal M, Sarilar TD, Cakil Saglik A, Bilgin M, Aydemir O, Barsan Kaya T, Tanir HM, Tekin AN. The effect of drip versus intermittent feeding on splanchnic oxygenation in preterm infants with intrauterine growth restriction: a prospective randomized trial. Eur J Pediatr. 2023 Mar;182(3):1317-1328. doi: 10.1007/s00431-023-04810-x. Epub 2023 Jan 13. PMID 36637540